CLINICAL TRIAL: NCT03566004
Title: Performance of a Non-invasive Test for the Detection of Helicobacter Pylori and Its Resistance to Clarithromycin in Stool by Real-Time PCR Amplidiag H. Pylori + ClariR (Mobidiag)
Brief Title: Performances of a H. Pylori Stool PCR Test
Acronym: HEPYSTOOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HEPYSTOOL
Record Dates: First submitted 2018-02-27; First posted 2018-06-21 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-03

CONDITIONS: Helicobacter Pylori

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endoscoped patients (Other): Patients addressed for endoscopy with indication of biopsies for H. pylori detection will be enroled to provide stool specimen
  Interventions: Diagnostic Test: Stool specimen collection

INTERVENTIONS:
Diagnostic Test: Stool specimen collection — The stool specimen collection was performed at the hospital or at home using a disposable device to be placed on the toilet seat and an E-nat Tube sent by postal to the lab.

SUMMARY:
Performance of a non-invasive test for the detection of Helicobacter pylori and its resistance to clarithromycin in stool by Real-Time PCR Amplidiag H. pylori + ClariR (Mobidiag).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* indication of endoscopy with biopsies for H. pylori infection
* Free subject, without tutorship or curatorship or subordination
* Patients benefiting from a social security scheme or benefiting through a third party
* Consent informed and signed by the patient after clear and fair information about the study

Exclusion Criteria:

* Age <18 years
* Contraindications to fibroscopy (suspicion of oesophageal perforation)
* Antibiotic intake less than 4 weeks old
* Diarrheal patients during sampling
* Patients who do not benefit from a social security scheme or who do not benefit from it through a third party
* Persons enjoying enhanced protection, namely minors, pregnant women, breastfeeding, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social institution, adults under legal protection, and finally patients in emergency situation.
* Pregnant or lactating women, women of childbearing potential who do not have effective contraception (hormonal / mechanical: oral, injectable, transcutaneous, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total oophorectomy )

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Detection of H. pylori by culture or glmM real-time PCR | Day 2
Detection of H. pylori by culture or glmM real-time PCR | Day30
Detection of clarithromycin resistance by E-test or Scorpion PCR from gastric biopsies. | Day 2
Detection of clarithromycin resistance by E-test or Scorpion PCR from gastric biopsies. | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Christophe BURUCOA, Principal Investigator — Poitiers University Hospital
Locations (1):
- CHU DE Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No